CLINICAL TRIAL: NCT01526096
Title: Pilot Study T Cell Depletion in the Setting of Autologous Stem Cell Transplantation for Patients With Multiple Myeloma
Brief Title: Stem Cell Transplantation for Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-551-B
Record Dates: First submitted 2011-08-10; First posted 2012-02-03 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Granulocyte Colony-Stimulating Factor; plerixafor; Blood Component Removal; Melphalan; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Standard ASCT (Grp 1) (Active Comparator): Standard autologous stem cell transplantation (ASCT)
  Interventions: Drug: G-CSF; Drug: Plerixafor; Procedure: Apheresis; Drug: Melphalan; Procedure: Stem cell re-infusion
- Depletion of T-cells after ASCT (Grp 2) (Experimental): Standard ASCT followed by treatment with basiliximab to remove certain immune cells (called regulatory T-cells or Tregs) from the blood
  Interventions: Drug: G-CSF; Drug: Plerixafor; Procedure: Apheresis; Drug: Melphalan; Procedure: Stem cell re-infusion; Drug: Basiliximab
- Depletion of T-cells before ASCT(Grp 3) (Experimental): Blood collected for an ASCT will be processed using a special cell sorting machine (CliniMACS device) to remove Treg cells before the stem cells are infused back into the body during stem cell transplant.
  Interventions: Drug: G-CSF; Drug: Plerixafor; Procedure: Apheresis; Drug: Melphalan; Procedure: Stem cell re-infusion; Device: CliniMACS CD25 microbeads and cell sorter

INTERVENTIONS:
Drug: G-CSF — G-CSF will be self-administered shot daily for 4 days pre-transplant. Up to 8 doses of G-CSF may be given. G-CSF will also be administered once daily under the skin beginning 5 days after your stem cell infusion until your white blood cell count is high enough
Drug: Plerixafor — Plerixafor (self-administered shot)prior to the beginning of the stem cell collection. Up to 4 doses of plerixafor may be given.
Procedure: Apheresis — Stem cell collection begins on day 5 and can last up to 3 days depending on the number collected.
Drug: Melphalan — Melphalan chemotherapy 100mg/m2 for 2 days after your admission into the hospital for your ASCT procedure.
  Other Names: Alkeran
Procedure: Stem cell re-infusion — Stem cells are thawed and reinfused back into the body via a catheter in the vein.
Drug: Basiliximab — Basiliximab (20mg) given by IV infusion (through the vein) 20-30 minutes the day after ASCT.
  Other Names: Simulect
  Arms: Depletion of T-cells after ASCT (Grp 2)
Device: CliniMACS CD25 microbeads and cell sorter — The stem cells collected during apheresis will be counted and treated with CD25 microbeads and processed by a special device called a CliniMACs machine which removes the regulatory T cells from you stem cell product.
  Arms: Depletion of T-cells before ASCT(Grp 3)

SUMMARY:
The purpose of this study is to test whether regulatory T-cell reduction is possible and safe in myeloma subjects undergoing autologous stem cell transplantation (ASCT).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma of any subtype in any disease stage, providing that patient does not have smoldering myeloma.
* Patient must otherwise be a candidate for ASCT as determined by treating physician.
* No current CNS Myeloma at time of enrollment.
* Life expectancy greater than 12 weeks.
* Age greater than or equal to 21 and less than or equal to 70 years old.
* EGOG performance status less than or equal to 2.
* No cardiac, pulmonary, hepatic, or renal contraindications for high dose chemotherapy.
* HIV Negative.
* No active Hepatitis B or C.
* Patients must be able to provide written informed, consent.

Exclusion Criteria:

* Pregnant or nursing women. Women of child-bearing age must be tested for pregnancy.
* Use of systemic immunosuppressive medications, including corticosteroids, tacrolimus, mycophenolate mofetil, sirolimus or cyclosporine A.
* Psychiatric illness which may make compliance to the clinical protocol unmanageable or which may compromise the ability of the patient to give informed consent.
* Active autoimmune disease including but not limited to: rheumatoid arthritis inflammatory bowel disease, celiac disease, systemic lupus erythematosis, scleroderma or multiple sclerosis.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07-12 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Purity of ex vivo depleted regulatory T cells prior to autologous stem cell transplant (arm 3 only) | 1-3 days
  Percentage of CD4+CD25+ regulatory T cells following ex vivo depletion in arm 3 will be analyzed by flow cytometry and compared to a pre-CD25-depletion sample. The depletion of CD25+ cells among the entire CD4+ population is expected to reach 80% efficiency.
Timing and duration of regulatory T cell depletion and recovery following autologous stem cell transplant | 180 days
  Timing and duration of regulatory T cell depletion and recovery following in vivo or ex vivo (arms 2 and 3) CD25+ T cell depletion will be performed at pre-defined timepoints prior to and following autologous stem cell transplant by flow cytometry on peripheral blood samples and directly compared to the percentages of regulatory T cells (CD4+CD25+FoxP3+ or CD4+CD25+CD127-) present at the same timepoints in patients enrolled onto arm 1 in which no regulatory T cell depletion is performed.
Incidence of autologous graft-versus-host disease following in vivo or ex vivo regulatory T cell depletion | 180 days
  The indicence of autologous graft-versus-host disease, as assessed by the development of skin rash, diarrhea and/or liver function test abnormalities consistent with autologous graft-versus-host disease following CD25+ T cell depletion and autologous stem cell transplant compared with the incidence of autologous graft-versus-host disease in patients enrolled onto arm 1 in which no regulatory T cell depletion is performed.

SECONDARY OUTCOMES:
Kinetics of recovery of peripheral blood cellular elements | 180 days
  Time to recovery of neutrophils and platelets will be analyzed by daily complete blood counts following autologous stem cell transplant. Patients enrolled onto arms 2 and 3 (in vivo and ex vivo regulatory T cell depletion, respectively) will be directly compared to patients enrolled onto arm 1 in which no regulatory T cell depletion is performed.
Number of patients that experience a complete response following autologous stem cell transplant based upon the assigned study arm using International Myeloma Working Group definitions | 100 days
  The complete response rate following autologous stem cell transplant with or without regulatory T cell depletion will be analyzed and compared directly between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bishop, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Derman BA, Zha Y, Zimmerman TM, Malloy R, Jakubowiak A, Bishop MR, Kline J. Regulatory T-cell depletion in the setting of autologous stem cell transplantation for multiple myeloma: pilot study. J Immunother Cancer. 2020 Jan;8(1):e000286. doi: 10.1136/jitc-2019-000286. PMID 31940591